CLINICAL TRIAL: NCT02922010
Title: A Follow-Up Survey of Oral Hygiene and Health Outcomes of Women Enrolled in the "OHMOM" Clinical Trial at the University of Alabama Birmingham
Brief Title: A Follow-Up Survey of Oral Hygiene and Health Outcomes for Women Previously Enrolled in "OHMOM"
Acronym: OHBABY
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015108
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The objective of this study is to assess oral health, oral hygiene knowledge, and daily oral hygiene practices of women who participated in a randomized controlled trial (2011001) at University of Alabama Birmingham during the period 2012-2014. Additional objectives of the research include evaluation of possible cultural, biological or other mechanisms for outcomes observed in the OHMOM clinical trial, and oral health screening of children born to mothers during the study for the purposes of understanding possible multigenerational effects of oral hygiene education.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* sign an informed consent form and be given a copy
* be a former subject in study 2011001 at University of Alabama Birmingham with a live birth outcome from that study.

Exclusion Criteria:

* any medical condition requiring pre-medication prior to dental procedures
* any diseases or conditions that might interfere with the subject safely completing the study
* inability to undergo study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from the OHMOM study and offspring from that study (NCT01549587) at the University of Alabama Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingivitis Index | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Gerlach, DDS, MPH, Study Director — Procter and Gamble
Locations (1):
- Center for Women's Reproductive Health, Birmingham, Alabama, United States